CLINICAL TRIAL: NCT03881540
Title: The Efficacy of a Transcultural Diabetes Nutrition Algorithm (tDNA) Care on Weight Loss and Metabolic Outcomes in Patients With Overweight, Obesity and Type 2 Diabetes in an Outpatient Clinic Setting
Brief Title: Efficacy of tDNA Care on Weight Loss and Metabolic Outcomes in Patients With Overweight, Obesity and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Winnie Chee, Principal Investigator, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMU R 134/2014
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDNA-MI group (Active Comparator): Follow tDNA intervention and motivational interviewing counselling
  Interventions: Other: tDNA-MI group
- tDNA-CC group (Active Comparator): Follow tDNA intervention and conventional counselling
  Interventions: Other: tDNA-CC group
- UC group (Other): Follow a conventional diet with standard diabetes support and lifestyle education
  Interventions: Other: UC group

INTERVENTIONS:
Other: tDNA-MI group — tDNA care with structured low calorie meal plan of 1200-1500 kcal/day with conventional foods + 1-2 serving of diabetes specific meal replacements and motivational interviewing counseling. .
  Arms: tDNA-MI group
Other: tDNA-CC group — tDNA care with structured low calorie meal plan of 1200-1500 kcal/day with conventional foods + 1-2 serving of diabetes specific meal replacements+ 150 min/week of moderate intensity exercise + and conventional counselling.
  Arms: tDNA-CC group
Other: UC group — Meal plan of 1200-1500 kcal/day using conventional foods + 150 min/week of moderate intensity exercise + and conventional counselling
  Arms: UC group

SUMMARY:
The aim of this study was to investigate the effectiveness of structured lifestyle intervention following a transcultural diabetes nutrition algorithm (tDNA) care compared to usual diabetes care in patients with overweight, obesity and type 2 diabetes (T2D), receiving either the motivational interviewing counseling or conventional counselling technique in an outpatient clinic setting.

The hypothesis is weight loss and glycated haemoglobin (A1C) level will be improved in patients following the tDNA care compared to usual diabetes care and the improvements will be greater in those receiving motivational interviewing counseling than conventional counselling.

DETAILED DESCRIPTION:
The main objective of this study was to investigate the effectiveness of structured lifestyle intervention following a transcultural diabetes nutrition algorithm (tDNA) care compared to usual diabetes care in patients with overweight, obesity and type 2 diabetes (T2D), receiving either the motivational interviewing counseling or conventional counseling technique in an outpatient clinic setting.

The specific objectives are:

1. To compare changes in the primary outcomes (weight, body mass index and A1C) in patients receiving structured lifestyle intervention based on tDNA care compared to usual diabetes care in addition to receiving either the motivational interviewing counseling or conventional counselling techniques at baseline, 6 months and 12 months of intervention.
2. To compare changes in the secondary outcomes (waist circumference, percentage body fat, fasting plasma glucose, lipid profile, high sensitivity-C-Reactive Protein and blood pressure) in patients receiving structured lifestyle intervention based on tDNA care compared to usual diabetes care in addition to receiving either the motivational interviewing counseling or conventional counselling techniques at baseline, and 6 months of intervention.
3. To compare the changes in dietary intake, Weight Efficacy Lifestyle, exercise and physical activity in patients receiving structured lifestyle intervention based on tDNA care compared to usual diabetes care in addition to receiving either the motivational interviewing counseling or conventional counselling techniques at baseline, 6 months and 12 months of intervention.

Study Design: This is a prospective open-label randomized clinical trial conducted in patients with overweight, obesity and T2D in an outpatient clinic setting.

Study duration: This study was conducted for a period of 12 months consisting of 6 months of intervention phase followed by subsequent 6 months of follow up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus, requiring weight loss
2. Treated with oral hypoglycaemic medications and/or lifestyle modifications
3. Medications have been optimised with no changes in pharmacotherapy in the past three months
4. Aged between 30 to 65 years
5. BMI of >23 kg/m²
6. A1C between 7% to 9%
7. Failed to achieve HbA1c reduction in the past three months even after seeing a dietitian
8. Willing to comply with study procedures.

Exclusion Criteria:

1. Patients whom weight loss might not be safe
2. Patients diagnosed with type 1 diabetes mellitus and type 2 diabetes mellitus with basal or multiple insulin injections
3. Patients with weight loss exceeding 5 kg in the past three months
4. Patients with current use of medications/meal replacements for weight loss
5. Patients with cancer requiring treatment for the past five years, except of non-melanoma skin cancers or cancers that have been clearly cured
6. Patients with history of bariatric surgery, small bowel resection, or extensive bowel resection
7. Patients with cardiovascular disease (heart attack or procedure within past three months or participation in cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischaemic attacks in the past three months, or documented history of pulmonary embolus for the past six months)
8. Patients receiving chronic treatment with systemic corticosteroids. Use of hormone replacement therapy or oral contraceptives will not lead to exclusion.
9. Patients with renal disease with eGFR <60 ml/min (based on MDRD) or currently receiving dialysis
10. Patients with chronic alcoholism
11. Patients who are currently pregnant or nursing
12. Patients who plan to relocate where it does not permit full participation in the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 6 months, 12 months
  Anthropometry
Change in Glycated haemoglobin (A1C) | 6 months, 12 months
  Biochemical measure

SECONDARY OUTCOMES:
Change in percentage body fat | 6 months
  Body composition
Change in fasting blood glucose | 6 months
  Biochemical measure
Change in total cholesterol, LDL-C and HDL-C | 6 months
  Biochemical measure
Change in High sensitivity C-Reactive Protein (HsCRP) | 6 months
  Biochemical measure
Change in systolic and diastolic blood pressure | 6 months
  Metabolic outcome
Change in energy intake and macronutrients | 6 months, 12 months
  Dietary intake
Change in Weight Efficacy Lifestyle (WEL) scores | 6 months, 12 months
  Eating self efficacy scores ranging from total scores of 0-180, subscales of 0-36. Total scores is a sum of subscales. Higher scores are better.
Change in exercise minutes | 6 months, 12 months
  Exercise

CONTACTS AND LOCATIONS:
Overall Officials: Winnie SS Chee, PhD, Principal Investigator — IMU University, Malaysia
Locations (1):
- International Medical University, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilcharan Singh HK, Chee WSS, Hamdy O, Mechanick JI, Lee VKM, Barua A, Mohd Ali SZ, Hussein Z. Eating self-efficacy changes in individuals with type 2 diabetes following a structured lifestyle intervention based on the transcultural Diabetes Nutrition Algorithm (tDNA): A secondary analysis of a randomized controlled trial. PLoS One. 2020 Nov 30;15(11):e0242487. doi: 10.1371/journal.pone.0242487. eCollection 2020. PMID 33253259